CLINICAL TRIAL: NCT06867042
Title: A Double-blind, Randomized, Multicenter, Parallel, Placebo-controlled Clinical Study to Evaluate the Efficacy, Safety and Tolerability of Tacrolimus Lipid Suspension for Enema in Adult Subjects with Mild to Moderately Active Left-sided/Distal Ulcerative Colitis Who Had an Inadequate Response to the Treatment
Brief Title: Tacrolimus Lipid Suspension for Enema in Adult Subjects with Mild to Moderately Active Left-sided/Distal Ulcerative Colitis Who Had an Inadequate Response to the Treatment
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jina Pharmaceuticals Inc. (Industry)
Collaborators: Novum Pharmaceutical Research Services (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 72289801
Record Dates: First submitted 2025-03-05; First posted 2025-03-10 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Ulcerative Colitis (UC); Ulcerative Colitis, Active Moderate
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Enema

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tacrolimus Lipid Suspension for Enema (Experimental): Patients will be administered Tacrolimus (4 mg) Lipid Suspension for Enema via rectal route once daily for 28 days
  Interventions: Drug: Tacrolimus Lipid Suspension for enema
- Identical Tacrolimus-free Lipid Suspension for Enema (Placebo Comparator): Patients will be administered with identical Tacrolimus-free Lipid Suspension for Enema via rectal route once daily for 28 days
  Interventions: Drug: Identical Tacrolimus-free Lipid Suspension for Enema

INTERVENTIONS:
Drug: Tacrolimus Lipid Suspension for enema — Tacrolimus Lipid Suspension for enema 4 mg/vial
  Arms: Tacrolimus Lipid Suspension for Enema
Drug: Identical Tacrolimus-free Lipid Suspension for Enema — Identical Tacrolimus-free Lipid Suspension for Enema
  Arms: Identical Tacrolimus-free Lipid Suspension for Enema

SUMMARY:
The study will evaluate the effectiveness, safety and tolerability of tacrolimus lipid suspension for enema in adult patients with mild to moderately active ulcerative colitis who had an inadequate response or intolerance of at least 1 of aminosalicylates (5-ASAs), corticosteroids, azothiopurine, mercaptopurine and methotrexate and need an alternative therapy. There will be approximately 150 male and female subjects of 18 and 65 years of age enrolled. Patients will be randomized into two groups where Tacrolimus Lipid Suspension for Enema or Placebo (Tacrolimus-free) Lipid Suspension for Enema will be administered rectally once daily for 28 days.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients ≥ 18 years and ≤ 65 years of age.
2. Patients have a documented history of idiopathic ulcerative colitis based on standard endoscopic (colonoscopic) and histological criteria involving the whole or part of the left side of the colon [approximately 60 cm up from the anus (anal verge) to splenic flexure of colon], with mild to moderate active disease.
3. Patients with a score of at least 4 on the modified Mayo Score (mMS), including an endoscopy subscore of at least 2 and a rectal bleeding subscore of at least 1.
4. Patients who have inadequate response, loss of response, or intolerance of at least 1 of aminosalicylates (5-ASAs) (mesalamine, sulfasalazine, olsalazine, basalazide), corticosteroids, azothiopurine, mercaptopurine and methotrexate and need an alternative therapy as per the discretion of the Investigator.
5. Patients who have failed to achieve total resolution of all symptoms to topical and/or oral standard treatment regimen of aminosalicylates (mesalamine, sulfasalazine, olsalazine, basalazide) or corticosteroids, azathioprine, mercaptopurine and methotrexate over minimum 4-week duration and need an alternative therapy as per the discretion of the Investigator. Determination of the outcomes of prior therapies should be made after the completion of at least one induction regimen and one maintenance regimen, as appropriate, for the prior therapy.
6. The patients who do not show evidence of benefits with the use of Biologics (e.g. Anti-integrins, Anti-TNFalpha and Anti-interleukins) for ulcerative colitis can be enrolled in the study. However, after a washout duration of 5 half-lives from any prior biologic treatments prior to enrollment is required. A shorter washout duration (e.g., 3 half-lives) is acceptable if undetectable drug levels of the biologic can be demonstrated.

   Note: Absence of benefit (inadequate response) is defined as signs and symptoms of persistently active disease despite an adequate trial of induction treatment with an anti-TNF-α agent (per country's approved label); OR recurrence of symptoms during maintenance dosing following prior clinical benefit;
7. A female participant is eligible to participate if she is not pregnant or breastfeeding, and at least one of the following conditions applies:

   1. Is not a woman of childbearing potential (WOCBP) OR
   2. Is a WOCBP and agrees to remain on an acceptable contraceptive method that is highly effective (with a failure rate of <1% per year), preferably with low user dependency when used consistently and correctly during the intervention period and for at least 6 weeks after the last dose of study intervention. The investigator should evaluate the effectiveness and the potential for contraceptive method failure (e.g., noncompliance, recently initiated) of the contraceptive method in relationship to the first dose of study intervention.
   3. A WOCBP must have a negative pregnancy test (serum) at screening and a negative pregnancy test (urine) before the first dose of study intervention.

   Note: The investigator is responsible for review of medical history, menstrual history, and recent sexual activity to decrease the risk for inclusion of a woman with an early undetected pregnancy.
8. Male participants are eligible to participate if they agree to the following during the intervention period and for at least 6 weeks after the last dose of study intervention:

   1. Must agree not to donate sperm for the purpose of reproduction

      PLUS EITHER OF B or C:
   2. Be abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long-term and persistent basis) and agree to remain abstinent OR
   3. Must agree to use contraception /barrier as detailed below

   i. A male participant must wear a condom when engaging in any activity that allows for passage of ejaculate to another person.

   ii. Male participants should also be advised of the benefit for a female partner to use a highly effective method of contraception as condom may break or leak when having sexual intercourse with a woman of childbearing potential who is not currently pregnant
9. Patient can understand and sign a written informed consent form, which must be obtained prior to initiation of study procedures.
10. Patients with adequate vitals, hematologic, liver and renal function at screening visit
11. If drugs such as aminosalicylates (e.g., mesalamine, sulfasalazine, olsalazine, balsalazide) or corticosteroids, azothiopurine, mercaptopurine and methotrexate recently discontinued, they must have been stopped for at least 2 weeks (for aminosalicylates, and corticosteroids)/8-week duration (for azathioprine, mercaptopurine, and methotrexate) prior to the endoscopy used for baseline modified Mayo Score (mMS).
12. For 30 patients undergoing intensive PK substudy:

    * Agree to undergo PK sampling procedure.
    * Participant having adequate venous access.

Exclusion Criteria:

1. Documented history of proximal or universal ulcerative colitis (pan colitis).
2. Patients who receive mMS score of 8 or greater (severe disease)
3. Patients with known allergy to study drugs or have a history of serious AEs related to their use.
4. Patients who demonstrate signs and symptoms of fulminant colitis, bowel stricture, toxic megacolon, an anticipated need for blood transfusion for gastrointestinal bleeding, or demonstrate evidence of peritonitis.
5. Prior documented history of high-grade dysplasia on biopsy from endoscopic examinations.
6. Presence of enteric pathogens or Clostridium difficile toxins in stool samples.
7. History of recurrent Clostridium difficile infection.
8. Patients who received systemic steroids or immunosuppressants within the previous 4 weeks of screening.
9. Treatment that included antibiotic, antifungal, or antiparasitic medications during screening.
10. Patients having a history of cancer (defined as malignancy), asthma, or bronchospasm.
11. Patients not able to withdraw from treatment or need continuing immunosuppressants for example sirolimus or cyclosporine during the study period.
12. Patients with hyperkalemia
13. Positive pregnancy test or lactating patients.
14. Patients with history or evidence of chemical substance abuse.
15. Patients with a history of failure to retain enemas.
16. Patients with Crohn's disease.
17. Patients with HIV, Hepatitis B and Hepatitis C infection
18. Patients who are currently using potassium sparing diuretics
19. Patients with pre-existent renal function disorders, liver function disorders, cardiac disease, hypertension, clinically important hematological, metabolic, psychiatric, central nervous system (CNS) or pulmonary disease.
20. Patients who participated in any other clinical or post-marketing study (not only for study drugs but also for medical devices) 30 days before signing the informed consent.
21. Any condition which the Investigator judges to preclude safe participation in the study or to confound the evaluation of the study outcome.
22. Uncontrolled hypertension (defined as systolic ≥140 mmHg or diastolic ≥90 mmHg) despite optimal antihypertensive treatment at screening. If blood pressure is out of range, up to 2 repeated assessments are permitted no more than 60 minutes apart.
23. Patient with severe hepatic impairment, defined as Child Pugh Class C.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients in clinical remission | Week 4
  Proportion of patients in clinical remission at week 4 will be calculated and reported. The difference between proportions of patients in clinical remission for test treatment and placebo and its 95% confidence interval will be calculated and reported